CLINICAL TRIAL: NCT06546436
Title: An Open, Dose-escalation Clinical Study to Evaluation of the Safety and Efficiency of a Single Dose of CARC-101C in Patients With Autoimmune Type 1 Diabetes Mellitus
Brief Title: The Safety and Efficiency of a Single Dose of CARC-101C in Patients With Autoimmune Type 1 Diabetes Mellitus
Status: Not yet recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School (Other)
Collaborators: Carcell Biopharma Ltd. (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Prevention
Other Study IDs: KMX-CARC-101C-IIT01
Record Dates: First submitted 2024-07-14; First posted 2024-08-09 (Actual); Last update posted 2024-08-09 (Actual); Status verified 2024-06

CONDITIONS: Autoimmune Type 1 Diabetes Mellitus(T1DM)

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Low-dose group (Active Comparator): Subjects enrolled in this group will received a one-dose injection of CARC-101C, 3×1010 eRBC(engineered Red Blood Cells) in one dose.
  Interventions: Drug: CARC-101C
- High-dose group (Active Comparator): Subjects enrolled in this group will received a one-dose injection of CARC-101C, 3×1011 eRBC in one dose.
  Interventions: Drug: CARC-101C

INTERVENTIONS:
Drug: CARC-101C — Subjects enrolled in the project will received a one-dose injection of CARC-101C

SUMMARY:
This study investigated the safety, efficiency, pharmacokinetics and pharmacokinetics of CARC-101C in patients with autoimmune type 1 diabetes. A single dose, dose escalation, open study design was used.

ELIGIBILITY:
Inclusion Criteria:

* Patients are eligible to be included in this study only if all of the following criteria apply:

  1. Males and females aged between ≥18 and ≤40 years old at the time of screening.
  2. Diagnosed with Autoimmune type 1 diabetes(T1D) within 3 to 6 months before screening, based on the 2021 version of the Chinese Guidelines for Diagnosis and Treatment of Type 1 Diabetes, with positive pancreatic autoantibodies:

     1. Must be tested Insulin a(utoantibody)IAA-positive at the time of diagnosis.
     2. Must not have undergone any form of insulin therapy before diagnosis.
  3. Currently undergoing insulin therapy and possesses HbA1c levels between ≥7.0% and ≤12%.
  4. Possess a body mass index (BMI) between at the time of screening ≥18.0 kg/m2 and ≤ 35.0 kg/m2.
  5. Fasting C-peptide ≥0.10 nmol/L (0.30 ng/ml) or post-MMTT peak C-peptide ≥0.2 pmol/mL (0.6 ng/mL).
  6. Males and females of childbearing potential must agree to use highly effective contraception, from providing informed consent till withdrawal or 3 months post-medication (whichever occurs later).
  7. Must be capable of providing written, signed, and dated informed consent and willing to comply with research requirements in the study.

Exclusion Criteria:

* Inclusion Criteria

Patients are eligible to be included in this study only if all of the following criteria apply:

1. Males and females aged between ≥18 and ≤40 years old at the time of screening.
2. Diagnosed with T1D within 3 to 6 months before screening, based on the 2021 version of the Chinese Guidelines for Diagnosis and Treatment of Type 1 Diabetes, with positive pancreatic autoantibodies:

   1. Must be tested IAA-positive at the time of diagnosis.
   2. Must not have undergone any form of insulin therapy before diagnosis.
3. Currently undergoing insulin therapy and possesses HbA1c levels between ≥7.0% and ≤12%.
4. Possess a body mass index (BMI) between at the time of screening ≥18.0 kg/m2 and ≤ 35.0 kg/m2.
5. Fasting C-peptide ≥0.10 nmol/L (0.30 ng/ml) or post-MMTT peak C-peptide ≥0.2 pmol/mL (0.6 ng/mL).
6. Males and females of childbearing potential must agree to use highly effective contraception, from providing informed consent till withdrawal or 3 months post-medication (whichever occurs later).
7. Must be capable of providing written, signed, and dated informed consent and willing to comply with research requirements in the study.

Exclusion Criteria

Patients are not eligible to be included in this study if any of the following criteria apply:

1. Average daily total insulin use was >1.0IU/kg(international unit) per day or <15IU per day 7 days before screening.
2. Any of the following abnormalities were detected in the laboratory during screening:

   1. Alanine aminotransferase (ALT) or aspartate aminotransferase (AST) >2 of ULN
   2. Total bilirubin >1.5 of ULN
   3. Hemoglobin <120g/L or > 165g/L (male), or < 110g/L or > 160g/L (female).
   4. Serum creatinine >1.5 of ULN(Upper limits of normal).
3. HIV-Ab or HBsAg or HCV-Ab(Hepatitis C virus) or treponema pallidum positive at screening
4. Have a serious/uncontrolled autoimmune disease in addition to T1D at the time of screening.
5. Have diabetic retinopathy stage 3 or above in addition requiring laser or surgical procedures 3 months prior to screening.
6. Possess pre-existing diseases affecting erythrocyte production and stability, including glucose-6-phosphate dehydrogenase (G6PD) deficiency, autoimmune hemolytic anemia, paroxysmal sleep hemoglobinuria, hereditary spherocytosis, hemoglobinopathy, pyruvate kinase deficiency etc.
7. History of acute or chronic pancreatitis.
8. History of hereditary bleeding tendency or coagulation dysfunction, or have a history of thrombosis, hemolysis or bleeding.
9. Diagnosed with DKA(Diabetic Ketoacidosis) or hyperosmotic hyperglycemia syndrome 1 month before screening.
10. Used immunosuppressants 3 months prior to screening.
11. Used systemic glucocorticoid therapy 2 weeks prior to screening or during the study period (except for inhaled and topical glucocorticoid therapies).
12. Participated in any drug or medical device clinical research within 3 months before screening.
13. Previously received cell therapy.
14. Previously reported malignant tumors (whether cured or not).
15. Systemic infection, severe trauma or other states of stress confirmed by laboratory tests or clinical manifestations at the time of screening.
16. Pregnant or lactating women.
17. Have other conditions that the investigator considers inappropriate to participate in this clinical study.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 12 (Estimated)
Dates: Start 2024-08-15 (Estimated); Primary Completion 2025-11-15 (Estimated); Study Completion 2027-05-31 (Estimated)

PRIMARY OUTCOMES:
Incidence and severity of adverse events within 3 weeks after administration (NCI CTCAE V5.0). | 21 days

SECONDARY OUTCOMES:
Changes of AUC(Area Under Curve) compared with baseline fasting and MMTT-stimulated C-peptide at 4, 12, 24, 36, 52 and 76 weeks. | 4, 12, 24, 36, 52 and 76 weeks
Changes of C-peptide compared with baseline in fasting and 2h after MMTT(Mixed-meal tolerance test)-stimulated at 4, 12, 24, 36, 52 and 76 weeks. | 4, 12, 24, 36, 52 and 76 weeks
Percentage of subjects with HbA1c < 7% at 12, 24, 36, 52 and 76 weeks. | 12, 24, 36, 52 and 76 weeks
Diachronic change of HbA1c from baseline at 12, 24, 36, 52 and 76 weeks. | 12, 24, 36, 52 and 76 weeks
Percentage of subjects whose weekly mean insulin requirement decreased by 50% or more at 4, 12, 24, 36, 52 and 76 weeks. | 4, 12, 24, 36, 52 and 76 weeks
Diachronic change in weekly mean insulin requirement from baseline at 4, 12, 24, 36, 52 and 76 weeks. | 4, 12, 24, 36, 52 and 76 weeks
Homeostatic model assessment of β-cell function (HOMA-β) from baseline at 4, 12, 24, 36, 52 and 76 weeks. | 4, 12, 24, 36, 52 and 76 weeks
Time in Range (TIR, time of glucose readings at 3.9 to 10.0 mmol/L) changes from baseline in indicators associated with continuous glucose monitoring at 12, 24, 36, 52 and 76 weeks. | 12, 24, 36, 52 and 76 weeks
Percentage of subjects with TIR >70% from baseline by continuous glucose monitors compared with baseline at 12, 24, 36, 52 and 76 weeks; | 12, 24, 36, 52 and 76 weeks
Maximum concentration observed (Cmax) of CARC-101C at Day1，Day2，Day5，Day7，Day21，Week4，Week12; | Day1，Day2，Day5，Day7，Day21，Week4，Week12
Time at which the maximum concentration (Tmax ) of CARC-101C at Day1，Day2，Day5，Day7，Day21，Week4，Week12; | Day1，Day2，Day5，Day7，Day21，Week4，Week12
AUC up to the last measurable concentratio（AUC (0-t)）: of CARC-101C at Day1，Day2，Day5，Day7，Day21，Week4，Week12; | Day1，Day2，Day5，Day7，Day21，Week4，Week12
AUC curve to infinite time（AUC (0--∞)） of CARC-101C at Day1，Day2，Day5，Day7，Day21，Week4，Week12; | Day1，Day2，Day5，Day7，Day21，Week4，Week12
Terminal phase rate constant(λz) of CARC-101C at Day1，Day2，Day5，Day7，Day21，Week4，Week12; | Day1，Day2，Day5，Day7，Day21，Week4，Week12
Terminal phase half-life (t1/2) of CARC-101C at Day1，Day2，Day5，Day7，Day21，Week4，Week12; | Day1，Day2，Day5，Day7，Day21，Week4，Week12
Changes of the T cell subpopulation compared with baseline at 3, 4, 12, 24, 36, 52 and 76 weeks; | 3, 4, 12, 24, 36, 52 and 76 weeks
Changes of the presence of pathogenicity related T cells compared with baseline at 3, 4, 12, 24, 36, 52 and 76 weeks; | 3, 4, 12, 24, 36, 52 and 76 weeks
Incidence and severity of adverse events within 76 weeks after administration according to version 5.0 of NCI CTCAE. | 76 weeks
Changes of Insulin Autoimmune Antibodies(IAA）compared with baseline at 4, 12, 24, 36, 52 and 76 weeks; | 4, 12, 24, 36, 52 and 76 weeks
Changes in cytokine levels. | 76 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Division of Endocrinology, the Affiliated Drum Tower Hospital of Nanjing University, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: Undecided